CLINICAL TRIAL: NCT06053112
Title: Safety and Efficacy of Infant Formula Containing a Specific Blend of Six Human Milk Oligosaccharides: A Double-blind, Randomized, Controlled Trial
Brief Title: The Trial of a New Infant Formula in Healthy Term Chinese Infants
Acronym: HexaHMO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Junlebao Dairy Group Co., Ltd. (Industry)
Collaborators: Merieux NutriSciences (China) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: JLB-CH002
Record Dates: First submitted 2023-06-26; First posted 2023-09-25 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Healthy Infants
Keywords: infant formula; HMOs

STUDY DESIGN:
Intervention Model Description: Test group: infant formula with 6 HMOs blend; Control group: infant formula without 6 HMOs blends
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Test group (Experimental): New infant formula with 6 HMOs blend
  Interventions: Other: New infant formula with 6 HMOs blend
- Control group (Active Comparator): Standard infant formula without 6 HMOs blend
  Interventions: Other: Standard infant formula without 6 HMOs blend
- Reference group (No Intervention): Breastfeeding

INTERVENTIONS:
Other: New infant formula with 6 HMOs blend — Infants are fed with HMO formula from the date of enrollment to the age of 6 months, exclusive formula feeding until the age of 4 months.
  Arms: Test group
Other: Standard infant formula without 6 HMOs blend — Infants are fed with standard formula from the date of enrollment to the age of 6 months, exclusive formula feeding until the age of 4 months.
  Arms: Control group

SUMMARY:
The aim of this randomized, controlled, multi-center, double-blind study of healthy term infants is to test the safety and efficacy of a new infant formula with a specific blend of six human milk oligosaccharides. The primary objective of the trial is to demonstrate the safety of the new infant formula supplemented by comparing the growth of infants randomized to the experimental formula versus the control formula from enrollment to the age of 4 months. The study has an interventional phase up to 6 months of age including 5 visits followed by an observational phase up to 12 months of age for a subgroup of the first 50 breastfed infants and the first 110 formula-fed infants including 2 additional visits.

ELIGIBILITY:
Inclusion Criteria:

1. Evidence of personally signed and dated informed consent indicating that the infant's both parents/legally acceptable representative(s) (LAR(s)), as per local regulation, have been informed of all pertinent aspects of the study.
2. Parents/LAR(s) of infants have reached the legal age of majority in China.
3. Parents/LAR(s) of infants are willing and able to comply with scheduled visits, and the requirements of the study protocol and can be contacted directly by telephone throughout the study.
4. At enrollment visit, infant post-natal age is ≤14 days (date of birth = day 0)
5. Healthy term infant (≥37 weeks of gestation).
6. Infant birth weight was ≥2500g and ≤4000g.
7. For formula-fed groups, infant is exclusively consuming and tolerating a cow' s milk infant formula since at least 3 days prior to enrollment. Its parents/LAR(s) have independently elected not to breastfeed.
8. For the breastfed REFERENCE group, infant has been exclusively consuming breastmilk since birth (small amounts of other feedings allowed during the first three days of life before breastfeeding is well-established), and its parents/LAR(s) have made the decision to continue exclusively breastfeeding until at least 4 months of age.

Exclusion Criteria:

1. Conditions requiring infant feedings other than those specified in the protocol.
2. Medical condition or history that could increase the risk associated with study participation or interfere with the interpretation of study results, including:

   * Evidence of major congenital malformations (e.g., cleft palate, extremity malformation).
   * Suspected or documented systemic or congenital infections (e.g., human immunodeficiency virus, cytomegalovirus, syphilis).
   * Previous or ongoing severe medical or laboratory abnormality (acute or chronic) which, in the judgment of the investigators, would make the infant inappropriate for entry into the study. Of note, infants who are normally healthy but at the time of enrollment suffering from acute illness in a minor condition which are common in infancy and do not require some of the exclusionary medication mentioned below can be enrolled.
3. Presently receiving or have received prior to enrollment any medication(s) or supplement(s) which are known or suspected to affect the following: fat digestion, absorption, and/or metabolism (e.g., pancreatic enzymes); stool characteristics and gut microbiota (e.g., oral, or systemic antibiotics, glycerine suppositories, bismuth-containing medications, docusate, Maltsupex, or lactulose); growth (e.g., insulin or growth hormone); gastric acid secretion.
4. Currently participating or having participated in another interventional clinical trial since birth.

Max Age: 14 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 326 (Estimated)
Dates: Start 2023-11-12 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Weight gain (g/day) between enrollment and the age of 4 months | until the age of 4 months

SECONDARY OUTCOMES:
Fecal secretory IgA (mg/g dry feces) at the age of 4 months corrected for baseline values | until the age of 4 months
Weight (g) at the ages of 42 days, 3 months, 4 months, 6 months and 12 months respectively | until the age of 12 months
Body length (cm) at the ages of 42 days, 3 months, 4 months, 6 months and 12 months respectively | until the age of 12 months
Body length gain (cm/week) at the ages of 42 days, 3 months, 4 months, 6 months and 12 months respectively | until the age of 12 months
Head circumference (cm) at the ages of 42 days, 3 months, 4 months, 6 months and 12 months respectively | until the age of 12 months
Head circumference gain (cm/week) at the ages of 42 days, 3 months, 4 months, 6 months and 12 months respectively | until the age of 12 months
Weight-for-age WHO growth standard z-scores at the ages of 42 days, 3 months, 4 months, 6 months and 12 months respectively | until the age of 12 months
Length-for-age WHO growth standard z-scores at the ages of 42 days, 3 months, 4 months, 6 months and 12 months respectively | until the age of 12 months
Weight-for-length WHO growth standard z-scores at the ages of 42 days, 3 months, 4 months, 6 months and 12 months respectively | until the age of 12 months
Head-circumference-for-age WHO growth standard z-scores at the ages of 42 days, 3 months, 4 months, 6 months and 12 months respectively | until the age of 12 months
Weight gain (g/day) between enrollment and the age of 6 months and 12 months respectively | until the age of 12 months
Stool pattern, GI symptoms and GI-related behaviors recorded in the retrospective 1-day questionnaire at baseline and in the prospective 3-day GI Symptom and Behavior Diary for 3 days prior to the age of 42 days, 3 months, 4 months, 6 months | until the age of 6 months
Fecal microbiome composition, diversity, community type assessed by NGS sequencing at baseline, the age of 4 months, 6 months and 12 months respectively | until the age of 12 months
Fecal acetic acid, propionic acid, butyric acid, isobutyric acid, valeric acid, isovaleric acid, and total short chain fatty acids at baseline, the age of 4 months, 6 months and 12 months respectively | until the age of 12 months
Fecal pH at baseline, the age of 4 months, 6 months and 12 months respectively | until the age of 12 months
Fecal secretory IgA (mg/g dry feces) at the age of 6 months corrected for baseline values | until the age of 6 months

OTHER OUTCOMES:
Faecal markers of immune health and gut inflammation and barrier integrity at baseline, the age of 4 months, 6 months and 12 months respectively | until the age of 12 months
  calprotectin, α-1-antitrypsin, lipocalin-2, claudin-3, cathelicidin, α-defensin and β-defensin assessed by ELISA
Illnesses and infections based on standard AE/SAE reporting | until the age of 12 months
Medication use based on standard AE/SAE reporting | until the age of 12 months
Breastmilk composition assessed by HPLC at baseline, the age of 42 days, 4 months and 6 months respectively | until the age of 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Wei CAI, MD, Ph.D., Principal Investigator — Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Locations (5):
- China (5):
  - Affiliated Hospital of Jining Medical College, Jining
  - Shanghai Public Health Clinical Center affiliated to Fudan University, Shanghai
  - Xinhua Hospital affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai
  - The Third People's Hospital affiliated to Hebei Medical University, Shijiazhuang
  - The First Teaching Hospital of Tianjin University of Traditional Chinese Medicine, Tianjin

IPD SHARING:
Plan to Share IPD: No